CLINICAL TRIAL: NCT06115109
Title: Observational Study, Prospective Multicentric, From the Natural History of Patients With Angelman Syndrome in Spain
Brief Title: Angelman Natural History Study - FAST Spain
Status: Recruiting | Type: Observational
Sponsor: Puerta de Hierro University Hospital (Other)
Collaborators: Parc Taulí Hospital Universitari (Other)
Responsible Party: Principal Investigator, BELEN RUIZ-ANTORAN, Principal Investigator, Puerta de Hierro University Hospital
Other Study IDs: 01_FAST SPAIN
Record Dates: First submitted 2022-07-26; First posted 2023-11-02 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Angelman Syndrome
MeSH Terms: conditions — Angelman Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non intervention, Observational study — Non intervention, Observational study

SUMMARY:
The goal of this study is to conduct a prospective, longitudinal study to observe the natural clinical progression and disease outcome of AS patients receiving no disease-modified intervention, with the purpose of obtaining data that will be useful for future clinical trials.

DETAILED DESCRIPTION:
The overall goal is to increase our understanding of the long-term natural history of Angelman syndrome and to identify and validate objective and sensitive outcome measures, which could serve as endpoints for outcome measures that can be used in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 3 months and 99 years of age.
2. Clinical diagnosis of Angelman Syndrome and molecular confirmation of the diagnosis.
3. The participant has an acceptable guardian capable of giving consent on behalf of the participant,
4. Willingness and ability of their guardians to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

1. Patients with any comorbidity that, in the clinical judgment of the principal investigator, may affect the results of the study. Any confirmed chronic or acute condition or illness affecting any system(s) that could interfere with study results and/or compliance with study procedures is included.
2. Patients who are participating in parallel studies with investigational drugs.
3. Unwillingness or inability of their guardians to follow the procedures outlined in the protocol.

Ages: 3 Months to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with a molecular diagnosis of Angelman syndrome
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Global Impression Scale for AS (CGI-AS) | 2 years
  Medical and neurological evaluation:
  -Clinical Global Impression Scale for AS (CGI-AS). The scale consists of several categories, from "not assessed" to "extremely severe." Professionals assess various aspects of behavior, communication, and the individual's overall functioning to assign a score on the CGI-AS scale. A higher score indicates a greater severity of symptoms, while a lower score indicates less severity.
Hammersmith Neonatal Neurological Examination (HINE) (for 0-2 years) | 2 years
  Medical and neurological evaluation:
  Hammersmith Neonatal Neurological Examination (HINE). 26 items that assess neurological function (cranial nerve function, posture, movements, tone, reflexes, and reactions). For neurological function, each item is individually scored on a scale of 0 to 3 based on descriptions and illustrative diagrams, so the total score can range from a minimum of 0 to a maximum of 78.

SECONDARY OUTCOMES:
Movement through actimetry | 2 years
  Continuous monitoring of movement through actimetry. Actigraphs will we placed on the non-dominant wrist or ankle of each participant. The motionlogger measures long-term gross motor activity and integrates degree and intensity of motion, and contains an accelerometer capable of sensing any motion with minimal resultant force of .01g. Actigraphy measurements will we recorded by the motionlogger every second using the proportional integrating measurement (PIM) mode of operation. In PIM mode, a numeric scale of movement activity is provided based on the absolute value of the area under the sensor curve. The PIM data can range from zero, corresponding to no movement when the limb is at rest, to a maximum value of 32,000, corresponding to the most vigorous and extreme movement of the limb.
Motor function scales | 2 years
  Motor function scales:
  - Functional Mobility Scale (FMS). The FMS classifies the functional mobility of children 4-18 years of age taking into account the assistive devices a child might use.
  3 items (distances), each of which is rated from 1-6 depending on assistance required, or "C" for crawling or "N" if distance is not completed Maximum score is a 6 for each of the distances (5m, 50m, and 500m)
Global development: Bayley Scale-3 (BSID-3) | 2 years
  -Bayley Scale-3 (BSID-3), at the time that version 4 of the Bayley scale (BSID-4) is validated in Spanish, it will be used in the context of the registry.
  Bayley Scales of Infant Development III, cognitive scale; raw scores used to reflect change over time and absolute growth (rather than standard scores) Range: Minimum =20 points; Maximum=60 Higher score = better outcome
Global development: Vineland Scale-III (VABS-III) | 2 years
  Vineland Scale-III is designed to measure adaptive behavior of individuals from birth to age 90. The Vineland-II contains 5 domains each with 2-3 subdomains. The main domains are: Communication, Daily Living Skills, Socialization, Motor Skills, and Maladaptive Behavior.
Global development: Aberrant behavior scale (ABC-C) | 2 years
  Aberrant behavior scale (ABC-C). The ABC-C is a global behavior checklist that measures drug and other treatment effects in people with developmental disabilities. It is made up of five subscales, including Irritability, Lethargy, Inappropriate Speech, Hyperactivity, and Stereotypy based on 58 items that describe various behavioral problems.
Communication assessment: ORCA communication tool (specifically designed for patients with AS) | 2 years
  ORCA communication tool (specifically designed for patients with AS). Observed Reported Communication Assessment (ORCA) Tool. Questionnaire designed to be completed by the patients' main carer and records patient communication.
Communication assessment: Leiter-3, Nonverbal Intelligence Scale | 2 years
  -Leiter-3, Nonverbal Intelligence Scale (for patients with equivalent developmental age greater than 3 years 6 months). Is a totally nonverbal test of intelligence and cognitive abilities. Evaluates nonverbal cognitive, attentional, and neuropsychological abilities, and targets 'typical' as well as 'atypical' children, adolescents, and now adults.
Sleep Disorders: Childhood Sleep Disorders Scale (Bruni Scale) | 2 years
  -Childhood Sleep Disorders Scale (Bruni Scale). The SDSC is a 26-item scale developed to assess the presence of sleep difficulties in children within the previous six months.
  Divided items into six categories representing some of the most common sleep diffi culties affecting adolescents and children: disorders of initiating and maintaining sleep, sleep breathing disorders, disorders of arousal/nightmares, sleep-wake transition disorders, disorders of excessive somnolence, and sleep hyperhidrosis (nighttime sweating).
  The measure is completed by the parent of the child and takes approximately 5-10 min to complete. Item 1 measures the child's average hours of sleep, from 1 ('9 - 11 h') to 5 ('less than 5 h'). Item 2 measures the child's average time to fall asleep, from 1 ('less than 15 min') to 5 ('more than 60 min'). The remaining 24 items are rated on a 5-point Likert scale, from 1 ('Never') to 5 ('Always [daily]').
Sleep Disorders: Children's Sleep Habits Questionnaire (CSHQ) | 2 years
  -Children's Sleep Habits Questionnaire (CSHQ) This questionnaire was designed as a sleep screening instrument for school-aged children that yields final scores across eight subscales: bedtime resistance, sleep resistance, parasomnia, sleep disordered breathing, night-wakings, daytime sleepiness, sleep anxiety, and sleep onset delay, as well as a summative score, called the Total Sleep Disturbance score.
Sleep Disorders: Diaries | 2 years
  This study will utilize a brief 6-item sleep diary to collect parent-reported sleep variables (e.g., "what time was your child down for the night?").
Proteomic analysis | 2 years
  Proteomic analysis: Ubiquitin proteomics approach. Characterization of ubiquitination by Ube3a, a proteasomal component conserved from yeast (Ddi1) to humans (DDI1 and DDI2).
Electroencephalogram (EEG) activity recordings | 2 years
  Electroencephalogram (EEG) to record brain activity of Angelman Syndrome patients over a 4-hour period (e.g., sleep architecture, number and frequency of seizures, background epileptic activity, delta-rhythmicity)

CONTACTS AND LOCATIONS:
Overall Officials: BELEN RUIZ ANTORAN, MD, Ph, Principal Investigator — Clinical Pharmacology Deparment, Hospital Universitario Puerta de Hierro Majadahonda
Locations (2):
- Spain (2):
  - Hospital Parc Tauli. Servicio de Genética molecular, Barcelona
  - Servicio de Farmacología Clínica. Hospital Universitario Puerta de Hierro Majadahonda, Madrid

IPD SHARING:
Plan to Share IPD: Undecided